CLINICAL TRIAL: NCT02656381
Title: Uveitis/Intraocular Inflammatory Disease Biobank (iBank)
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160046; 16-EI-0046
Record Dates: First submitted 2016-01-13; First posted 2016-01-14 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09-10

CONDITIONS: Uveitis
Keywords: Sarcoidosis; Behcet's Disease; Natural History Study; Biological Specimens; Immune System; Natural History
MeSH Terms: conditions — Uveitis; Sarcoidosis; Behcet Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Anterior Uveitis: Participants with AU at entry
- Intermediate Uveitis: Participants with IU at entry
- Other: Participants not fitting above criteria
- Posterior/Pan Uveitis: Participants with non-infectious posterior or pan-uveitis

SUMMARY:
Background:

Uveitis is a serious eye disease that can cause vision loss. Treatment sometimes causes serious side effects or does not work. Researchers want to learn more about uveitis and why some people develop it.

Objective:

To learn clinical and genetic factors that may make people develop uveitis and influence how they respond to treatment.

Eligibility:

People ages 8 and older who have uveitis, scleritis, inflammatory eye disease, or a disease related to eye inflammation

INCLUSION CRITERIA FOR COVID-19 COHORT:

Participants with COVID-19 will be eligible if they:

1. Have a diagnosis of COVID-19 confirmed by a nasaopharyngeal swab (or another confirmative test) within less than or equal to 3 days prior, with symptoms of any severity.
2. Are able to give verbal consent.
3. Are 16 years of age or older.

EXCLUSION CRITERIA FOR COVID-19 COHORT:

Participants with COVID-19 will not be eligible if they:

1. Use regular prescription eye drops on the day of sampling.
2. Current use of antiviral medications.

Design:

Participants will be screened with:

Medical history

Physical exam

Eye exam

Participation lasts up to 10 years. The clinic visit schedule varies depending on participants eye disease:

Baseline visit with annual follow-ups

Baseline visit, visits at months 3 and 6, and annual follow-ups

Another schedule set by the researcher

Depending on participants eye disease, tests during each visit could include:

Fluorescein angiography or indocyanine green angiography: Dye is injected through a needle in the arm

and flows through the blood vessels in the eye. A camera takes pictures of the eye.

Electroretinography: Participants sit in the dark with their eyes patched.

After 30 minutes, numbing drops and contact lenses are put in the eyes. Then, the retina is stimulated with flashing lights.

Perimetry: Participants look into a bowl or lens and press a button when they see a light.

Conjunctival or corneal biopsy, or skin biopsy: A small piece of tissue is removed.

Anterior chamber tap: A needle enters the eye to remove fluid.

Blood and urine tests

Saliva, stool, hair, or tear samples

Cotton swab of the inside of the cheek.

During the study, participants may need immunosuppressive treatment, such as drugs or injections in or around the eyes depending on their disease.

DETAILED DESCRIPTION:
Uveitis refers to a large group of intraocular inflammatory diseases that can cause devastating visual loss in adults and children. This study establishes a clinical database and biospecimen repository for the identification of novel factors relevant to the pathogenesis, progression, and response to treatment of a wide spectrum of uveitic conditions.

Objectives: This study provides for standardized collection of longitudinal clinical data and for serial collection, processing, and storage of a variety of biospecimens. The clinical data set and biospecimen repository will be used to identify novel genetic factors, biomarkers, and experimental models associated with pathogenesis, progression, and response to treatment for various ocular and systemic conditions where inflammation of the uveal tract is present.

Study Population: The study plans to accrue 550 participants with uveitis or related diseases. This will not be restricted by anatomical location or etiology with the inclusion of both idiopathic cases, infectious uveitis, scleritis and those cases linked to a disease known to be associated with an increased risk of intraocular inflammation (e.g., sarcoidosis, Beh(SqrRoot) (Beta)et's disease and multiple sclerosis (MS) and lymphoma). In addition, 100 participants without intraocular inflammatory disease will be enrolled as controls.

Design: This is a prospective observational study of participants with intraocular inflammatory diseases incorporating: 1. A standardized follow-up and testing schedule with standard-of-care management of eye diseases; and/or 2. Collection of biospecimens for research purposes for which sampling does not incur more than minimal risk to participants. Outcome Measures: Outcome measures include the interaction of key parameters of disease phenotype (such as visual acuity and ocular imaging features) with genetic variants and other biomarkers identified from biospecimens and the characterization of new experimental models of eye health and disease.

ELIGIBILITY:
* INCLUSION CRITERIA (NOT APPLICABLE TO COVID COHORT):

Participants will be eligible if they:

1. Have a diagnosis of uveitis, scleritis or a disease known to be associated with intraocular inflammation, (e.g., sarcoidosis, Behcet's disease, MS and lymphoma) OR could serve as an unaffected control.
2. Are eight years of age or older if an affected participant.
3. Are 18 years of age or older if serving as an unaffected control.
4. For participants 18 years of age and older:

   * Are willing to give informed consent that includes collection and study of at least one peripheral blood sample.

EXCLUSION CRITERIA (NOT APPLICABLE TO COVID COHORT):

Participants will not be eligible if they:

1. Are unable to understand and sign the informed consent form.
2. Are unable or unwilling to give informed consent that includes use of medical records and clinical samples for current and future research related to vision and diseases affecting the eyes.
3. Have a systemic disease that compromises the ability to provide adequate ophthalmologic examination or treatment as determined by the investigator.
4. For participants with uveitis:

   * Have inactive anterior uveitis or quiescent infectious uveitis not requiring such regimented and intensive standardized testing as determined by the Investigator.
   * Have end stage or chronic quiescent changes in the setting of an established infectious etiology, such as an old ocular toxoplasma scar (participants with active intraocular inflammation due to infection will be recruited).

The eligibility requirements for this protocol are intended to be broadly inclusive, but those individuals screened at the NEI and found to be ineligible may be evaluated under the NEI Screening Protocol for potential participation in other studies.

INCLUSION CRITERIA FOR COVID-19 COHORT:

Participants with COVID-19 will be eligible if they:

1. Have a diagnosis of COVID-19 confirmed by a nasopharyngeal swab (or another confirmative test) within less than or equal to 3 days prior, with symptoms of any severity.
2. Are able to give verbal consent.
3. Are 16 years of age or older.

EXCLUSION CRITERIA FOR COVID-19 COHORT:

Participants with COVID-19 will not be eligible if they:

1. Use regular prescription eye drops on the day of sampling.
2. Current use of antiviral medications.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study plans to accrue 550 participants with uveitis or related diseases. This will not be restricted by anatomical location or etiology with the inclusion of both idiopathic cases, infectious uveitis, scleritis and those cases linked to a disease known to be associated with an increased risk of intraocular inflammation (e.g., sarcoidosis, Beh(SqrRoot)(Beta)et's disease, multiple sclerosis (MS) and lymphoma). In addition, 100 participants without intraocular inflammatory disease will be enrolled as controls.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
The clinical data and samples from this study will be used to test for interaction of key parameters of phenotype with genetic variants and other biomarkers identified from biospecimens. | 7 years
  The intent is to collect data on a variety of phenotypic pararmeters and to store biospecimens in a manner that permits a broad array of potnential testing and experimentation in the future.

SECONDARY OUTCOMES:
Secondary outcomes will include the number and severity of systemic and ocular adverse events among participants who use systemic immunosuppression. | 7 years
  Events include but are not limited to structural ocular complications, hospitalizations, osteoporosis, renal and hepatic side effects, infections and myelosuppression from conventional immunosuppressives and biologics

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei J, Mattapallil MJ, Horai R, Jittayasothorn Y, Modi AP, Sen HN, Gronert K, Caspi RR. A novel role for lipoxin A4 in driving a lymph node-eye axis that controls autoimmunity to the neuroretina. Elife. 2020 Mar 2;9:e51102. doi: 10.7554/eLife.51102. PMID 32118582
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-EI-0046.html